CLINICAL TRIAL: NCT04925752
Title: A Phase 3, Double-Blind, Multicenter, Randomized Study to Evaluate the Efficacy and Safety of Subcutaneous Twice Yearly Long-Acting Lenacapavir for HIV Pre-Exposure Prophylaxis in Cisgender Men, Transgender Women, Transgender Men, and Gender Nonbinary People ≥ 16 Years of Age Who Have Sex With Male Partners and Are at Risk for HIV Infection
Brief Title: Study of Lenacapavir for HIV Pre-Exposure Prophylaxis in People Who Are at Risk for HIV Infection
Acronym: PURPOSE 2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GS-US-528-9023; DOH-27-102021-6681 (Other: South African National Clinical Trial Registry)
Record Dates: First submitted 2021-05-28; First posted 2021-06-14 (Actual); Results first posted 2025-09-17 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Pre-Exposure Prophylaxis of HIV Infection
MeSH Terms: interventions — lenacapavir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; emtricitabine tenofovir alafenamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Randomized Blinded Phase: LEN + Placebo-to-match (PTM) F/TDF (Experimental): Participants will receive the following for up to approximately 52 weeks:
  * Subcutaneous (SC) lenacapavir (LEN) 927 mg every 26 weeks
  * Oral PTM Emtricitabine/Tenofovir Disoproxil Fumarate (F/TDF) once daily
  * Oral LEN 600 mg on Days 1 and 2
  Participants will receive oral LEN if SC injections are not available.
  Interventions: Drug: Oral Lenacapavir (LEN); Drug: Sub-cutaneous (SC) Lenacapavir (LEN); Drug: PTM F/TDF
- Randomized Blinded Phase: Placebo LEN + F/TDF (Experimental): Participants will receive the following for up to approximately 52 weeks:
  * SC LEN placebo every 26 weeks
  * Oral F/TDF 200/300 mg once daily
  * PTM Oral LEN on Days 1 and 2
  Participants will receive oral LEN placebo if SC injections are not available.
  Interventions: Drug: F/TDF; Drug: Placebo SC LEN; Drug: PTM Oral LEN
- LEN Open-Label Extension (OLE) Phase (Experimental): Participants will be offered entry into LEN OLE Phase, following completion of primary analysis, if LEN demonstrates acceptable safety and efficacy in the Randomized Blinded Phase.
  Participants randomized to LEN will continue to receive SC LEN 927 mg, every 26 weeks (± 7 days), and have study visits every 13 weeks (± 7 days).
  Participants randomized to F/TDF will switch to SC LEN 927 mg on OLE Day 1, Week 26 and every 26 weeks thereafter. Participants will also receive oral LEN 600 mg on OLE Days 1 and 2.
  All participants in LEN OLE Phase will complete the phase, once LEN becomes available or the sponsor decides to discontinue the study, whichever happens first.
  After completing LEN OLE Phase or study discontinuation, participants will transition to local PrEP, including LEN or other options. If a participant exits early, they will complete an early study drug discontinuation (ESDD), be referred to local PrEP services if needed, and have a 30-day follow-up visit.
  Interventions: Drug: Oral Lenacapavir (LEN); Drug: Sub-cutaneous (SC) Lenacapavir (LEN)
- Pharmacokinetic (PK) Tail Phase (Experimental): Participants who prematurely discontinue study drug during the Randomized Blinded Phase and participants that were randomized to LEN who choose not to continue in the LEN OLE Phase will transition to the PK Tail Phase. Participants will receive oral F/TDF (or Emtricitabine/Tenofovir Alafenamide (F/TAF) for US participants only) once daily for 78 weeks to cover the PK tail and complete visits every 13 weeks (+/- 7 days).
  Upon unblinding, participants who were randomized to F/TDF in the Randomized Blinded Phase who decline to participate in the LEN OLE Phase will complete the ESDD visit, transition to local HIV prevention services, and return for a 30-day follow-up visit.
  Interventions: Drug: F/TDF; Drug: F/TAF (for US participants only)

INTERVENTIONS:
Drug: Oral Lenacapavir (LEN) — Tablets administered orally without regard to food
  Other Names: GS-6207
  Arms: LEN Open-Label Extension (OLE) Phase; Randomized Blinded Phase: LEN + Placebo-to-match (PTM) F/TDF
Drug: F/TDF — Tablets administered orally
  Other Names: Truvada®
  Arms: Pharmacokinetic (PK) Tail Phase; Randomized Blinded Phase: Placebo LEN + F/TDF
Drug: Sub-cutaneous (SC) Lenacapavir (LEN) — Administered via SC injections
  Other Names: GS-6207; Yeztugo
  Arms: LEN Open-Label Extension (OLE) Phase; Randomized Blinded Phase: LEN + Placebo-to-match (PTM) F/TDF
Drug: Placebo SC LEN — Administered via SC injections
  Arms: Randomized Blinded Phase: Placebo LEN + F/TDF
Drug: PTM F/TDF — Tablets administered orally
  Arms: Randomized Blinded Phase: LEN + Placebo-to-match (PTM) F/TDF
Drug: PTM Oral LEN — Tablets administered orally
  Arms: Randomized Blinded Phase: Placebo LEN + F/TDF
Drug: F/TAF (for US participants only) — F/TAF tablets administered orally once daily
  Other Names: Descovy
  Arms: Pharmacokinetic (PK) Tail Phase

SUMMARY:
The goal of this study is to evaluate the efficacy of the study drugs, lenacapavir (LEN) in preventing HIV infection, in participants ≥ 16 years of age who have condomless receptive anal sex with partners assigned male at birth and are at risk for HIV-1 infection.

The primary objective of this study is to evaluate the efficacy of LEN for HIV-1 PrEP in participants ≥ 16 years of age who have condomless receptive anal sex with partners assigned male at birth at risk of HIV-1 infection.

ELIGIBILITY:
Key Inclusion Criteria:

Incidence Phase

* CGM, TGW, TGM, and GNB who have condomless receptive anal sex with partners assigned male at birth and are at risk for HIV infection.
* HIV-1 status unknown at screening and no prior HIV-1 testing within the last 3 months.
* Sexually active with ≥ 1 partner assigned male at birth (condomless receptive anal sex) in the last 12 months and 1 of the following:

  * Condomless receptive anal sex with ≥ 2 partners in the last 12 weeks.
  * History of syphilis, rectal gonorrhea, or rectal chlamydia in the last 24 weeks.
  * Self-reported use of stimulants with sex in the last 12 weeks.

Randomized Phase

* Negative local rapid fourth generation HIV-1/2 Ab/Ag, central fourth generation HIV-1/2 Ab/Ag, and HIV-1 RNA quantitative nucleic acid amplification testing (NAAT).
* Estimated glomerular filtration rate (eGFR) ≥ 60 mL/min at screening according to the Cockcroft-Gault formula for creatinine clearance (CLcr).

Key Exclusion Criteria:

Incidence Phase

* Prior use of HIV PrEP (including F/TDF or F/TAF) or HIV postexposure prophylaxis (PEP) in the past 12 weeks or any prior use of long-acting systemic PrEP (including cabotegravir or islatravir).
* Prior recipient of an HIV vaccine or HIV broadly neutralizing antibody formulation.

Randomized Phase

* Acute viral hepatitis A, B or C or evidence of chronic hepatitis B or C infection.
* Severe hepatic impairment or a history of or current clinical decompensated liver cirrhosis.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Cisgender male (CGM), Transgender male (TGM), Transgender women (TGW), and Gender non-binary (GNB)
Enrollment: 3292 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2028-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (93):
- United States (60):
  - UAB Sexual Health Research Clinic, Birmingham, Alabama
  - Loma Linda University Clinical Trial Center Clinic, Loma Linda, California
  - Ruane Clinical Research Group Inc., Los Angeles, California
  - UCLA CBAM Vine Street Clinic, Los Angeles, California
  - Charles R. Drew University of Medicine and Science (CDU) - Clinical Translational Research Center (CTRC), Los Angeles, California
  - Mills Clinical Research, Los Angeles, California
  - The Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Los Angeles, California
  - BIOS Clinical Research, Palm Springs, California
  - UCSD Anti Viral Research Center, San Diego, California
  - Bridge HIV at the San Francisco Department of Public Health, San Francisco, California
  - Optimus Medical Group, San Francisco, California
  - University of Colorado Clinical and Translational Research Centers (CTRC), Aurora, Colorado
  - Yale University, School of Medicine, New Haven, Connecticut
  - Whitman-Walker Institute Inc., Washington D.C., District of Columbia
  - Washington Health Institute, Washington D.C., District of Columbia
  - Therafirst Medical Center, Fort Lauderdale, Florida
  - Gary Richmond, MD, PA, Fort Lauderdale, Florida
  - Midway Immunology & Research Center, LLC, Ft. Pierce, Florida
  - CAN Community Health Clinic, Jacksonville, Florida
  - University of Miami Miller School of Medicine Division of Infectious Disease Research - Converge Miami, Miami, Florida
  - CAN Community Health, Miami Gardens, Florida
  - Orlando Immunology Center, Orlando, Florida
  - CAN Community Health, Sarasota, Florida
  - The Hope Clinic at Emory University, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Emory University Hospital Midtown Infectious Disease Clinic, Atlanta, Georgia
  - RMR Core Center, Chicago, Illinois
  - University of Illinois at Chicago, Department of Medicine, Division of Infectious Diseases, Project WISH, Chicago, Illinois
  - Howard Brown Health Center, Chicago, Illinois
  - Indiana University Infectious Diseases Research, Indianapolis, Indiana
  - Baptist Health Lexington, Lexington, Kentucky
  - Norton Infectious Disease Specialists, Louisville, Kentucky
  - LSU-CrescentCare Sexual Health Center- New Orleans Community Health Center, New Orleans, Louisiana
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - The Fenway Institute, Boston, Massachusetts
  - Be Well Medical Center, Berkley, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Open Arms Healthcare Center, Jackson, Mississippi
  - KC CARE Health Center, Kansas City, Missouri
  - St. Michael's Medical Center, Newark, New Jersey
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - Icahn School of Medicine at Mount Sinai- Mount Sinai Downtown, New York, New York
  - NC TraCS Institute - CTRC; University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cone Health/Regional Center for Infectious Disease Research Center, Greensboro, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Penn Prevention Unit, Philadelphia, Pennsylvania
  - Philadelphia FIGHT Community Health Centers, Jonathan Lax Treatment Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Infectious Disease Clinic, Charleston, South Carolina
  - Prisma Health-Midlands Clinical Research Unit, Columbia, South Carolina
  - Prisma Health Internal Medicine Clinic, Greenville, South Carolina
  - Methodist University Hospital/University of Tennessee Health Science Center, Clinical Research Center, Memphis, Tennessee
  - St Jude Children's Research Hospital, Memphis, Tennessee
  - Meharry Medical College Clinical and Transitional Research Center, Nashville, Tennessee
  - Central Texas Clinical Research, Austin, Texas
  - Centro San Vincente, El Paso, Texas
  - UT Health Science Center at Houston, Houston, Texas
  - The Crofoot Research Center, INC, Houston, Texas
  - Ofiice of Dr. Peter Shalit, MD, Seattle, Washington
- Argentina (3):
  - Hospital General de Agudos JM Ramos Mejia, Buenos Aires
  - Fundacion Huesped, Buenos Aires
  - Instituto de Investigaciones Clinicas Mar del Plata, Buenos Aires
- Brazil (9):
  - Unidade de Pesquisa Clinica em Vacinas (UPqVac) da Faculdade de Medicina da Universidade, Belo Horizonte - MG
  - Fundação Bahiana de Infectologia, Canela-Salvador
  - Fundação de Medicina Tropical Doutor Heitor Vieira Dourado / Fundação Medicina Tropical do Amazonas - FMT/IMT/AM, Manauas
  - Hospital General de Nova Iguaçu - HGNI, Nova Iguaçu
  - Grupo Hospitalar Conceição/ Hospital Nossa Senhora da Conceição S.A., Porto Alegre
  - Instituto Nacional de Infectologia Evandro Chagas / Fundação Oswaldo Cruz - INI FIOCRUZ, Rio de Janeiro
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo
  - Centro de Referência e Treinamento DST/AIDS, São Paulo
  - Center for Management and Research. SPDM-Paulista Association for the Development of Medicine-Hospital São Paulo/Federal, São Paulo
- Centro de Investigacion Farmaceutica Especializada de Occidente S.C., Guadalajara C.P., Mexico
- Peru (5):
  - Asociacion Civil Impacta Salud y Educacion - Sede Barranco, Barranco
  - Instituto de Medicina Tropical "Daniel Alcides Carrion", Facultad de Medicina Humana, UNMSM, Callao
  - Asociacion Civil Selva Amazonica, Iquitos
  - Via Libre, Lima
  - Asociacion Civil Impacta Salud y Educacion - Sede San Miguel, Lima
- Puerto Rico (2):
  - Ararat Research Center, San Juan, PR
  - Centro Ararat- San Juan, San Juan, PR
- South Africa (6):
  - Desmond Tutu Health Foundation, Cape Town
  - Wits Reproductive Health and HIV Institute (Wits RHI), Johannesburg
  - The Aurum Institute: Pretoria Clinical Research Centre, Pretoria
  - Setshaba Research Centre, Soshanguvhe
  - The Aurum Institute Tembisa CRC, Clinic 4, Tembisa
  - FPD-DTHF Ndevana Commuity Research Site, Vincent
- Thailand (7):
  - Institute of HIV Research and Innovation, Bangkok
  - King Chulalongkorn Memorial Hospital, Bangkok
  - The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT), Thai Red Cross AIDS research Centre, Bangkok
  - Ramathibodi Hospital, Mahidol University, Bangkok
  - Research Institute for Health Sciences, Chiang Mai University, Chiang Mai
  - Srinagarind Hospital, Khon Kaen University, Khon Kaen
  - Bamrasnaradura Infectious Disease Institute, Nonthaburi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kelley CF, Acevedo-Quiñones M, Agwu AL, et al. Twice-yearly lenacapavir PrEP in cisgender gay men, transgender women and men, and gender-diverse people (PURPOSE 2). Presented at: HIV Drug Therapy Glasgow; November 10-13, 2024; Glasgow, United Kingdom.
- [Background] Kelley CF, Acevedo-Quinones M, Agwu AL, Avihingsanon A, Benson P, Blumenthal J, Brinson C, Brites C, Cahn P, Cantos VD, Clark J, Clement M, Creticos C, Crofoot G, Diaz RS, Doblecki-Lewis S, Gallardo-Cartagena JA, Gaur A, Grinsztejn B, Hassler S, Hinojosa JC, Hodge T, Kaplan R, Lacerda M, LaMarca A, Losso MH, Valdez Madruga J, Mayer KH, Mills A, Mounzer K, Ndlovu N, Novak RM, Perez Rios A, Phanuphak N, Ramgopal M, Ruane PJ, Sanchez J, Santos B, Schine P, Schreibman T, Spencer LY, Van Gerwen OT, Vasconcelos R, Vasquez JG, Zwane Z, Cox S, Deaton C, Ebrahimi R, Wong P, Singh R, Brown LB, Carter CC, Das M, Baeten JM, Ogbuagu O; PURPOSE 2 Study Team. Twice-Yearly Lenacapavir for HIV Prevention in Men and Gender-Diverse Persons. N Engl J Med. 2025 Apr 3;392(13):1261-1276. doi: 10.1056/NEJMoa2411858. Epub 2024 Nov 27. PMID 39602624
- [Background] Cespedes M, Das M, Hojilla JC, Blumenthal J, Mounzer K, Ramgopal M, Hodge T, Torres TS, Peterson C, Shibase S, Elliott A, Demidont AC, Callaghan L, Watson CC, Carter C, Kintu A, Baeten JM, Ogbuagu O. Proactive strategies to optimize engagement of Black, Hispanic/Latinx, transgender, and nonbinary individuals in a trial of a novel agent for HIV pre-exposure prophylaxis (PrEP). PLoS One. 2022 Jun 3;17(6):e0267780. doi: 10.1371/journal.pone.0267780. eCollection 2022. PMID 35657826
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-528-9023

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4807 participants were screened. Out of 4807, 4634 participants had at least 1 non-missing HIV-1 diagnosis based on HIV test results from a central laboratory. Therefore, 4634 participants were considered for screening in the Incidence Phase and were included in the All Screened Set. Out of 4634, 3292 were enrolled and randomized in Randomized Blinded Phase. Incidence Phase refers to the Screening Phase.
Pre-assignment Details: Participants were enrolled in Argentina, Brazil, Mexico, Peru, South Africa, Thailand, Puerto Rico and United States. Data submitted represent primary analysis from data collected by Primary Completion Date (PCD) (Per pre-specified analysis, PCD is when at least 50% of the planned randomized participants were followed up for at least 52 weeks in the study or prematurely discontinued from the study). Complete data will be submitted within 1 year of actual study completion date.
Groups:
- Randomized Blinded Phase: LEN + Placebo-to-match (PTM) F/TDF: Participants received lenacapavir (LEN) 927 mg subcutaneous (SC) injection, every 26 weeks, starting on Day 1 for up to approximately 52 weeks. Participants also received loading dose of LEN 600 mg tablet orally, once daily on Day 1 and Day 2. Participants received placebo to match (PTM) emtricitabine/tenofovir disoproxil fumarate (F/TDF) tablet orally, once daily, up to approximately 52 weeks.
- Randomized Blinded Phase: Placebo LEN + F/TDF: Participants received F/TDF tablet on Day 1 orally, once daily for up to approximately 52 weeks. Participants also received PTM LEN SC injection every 26 weeks starting on Day 1 up to approximately 52 weeks and PTM LEN tablet, orally, once daily on Day 1 and Day 2.
Period: Overall Study
Arm/Group | Randomized Blinded Phase: LEN + Placebo-to-match (PTM) F/TDF | Randomized Blinded Phase: Placebo LEN + F/TDF
Started | 2195 | 1097
Completed (Completed = Discontinued and entered into Open-label F/TDF (or F/TAF for US participants only) Treatment Phase.) | 123 | 32
Not Completed | 2072 | 1065
Not completed — Still on Study | 1826 | 926
Not completed — Withdrew Consent | 128 | 59
Not completed — Lost to Follow-up | 73 | 47
Not completed — Randomized but Never Treated | 12 | 9
Not completed — Hiv-1 Infection | 6 | 7
Not completed — Investigator's discretion | 8 | 5
Not completed — Non-compliance with Study Drug | 8 | 5
Not completed — Adverse Event | 5 | 2
Not completed — Death | 4 | 2
Not completed — Protocol Violation | 1 | 3
Not completed — Withdrew Assent | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Randomized Blinded Phase Safety Analysis Set included all participants who took at least 1 dose of any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomized Blinded Phase: LEN + Placebo-to-match (PTM) F/TDF | Randomized Blinded Phase: Placebo LEN + F/TDF | Total
Number analyzed (Participants) | 2183 | 1088 | 3271
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (8.7) | 31 (9.5) | 30 (9.0)
Age, Customized [Count of Participants; unit: Participants]
  16 to <18 years | 3 | 1 | 4
  18 to ≤ 25 years | 749 | 343 | 1092
  > 25 to < 35 years | 912 | 423 | 1335
  35 to < 50 years | 454 | 267 | 721
  ≥ 50 years | 65 | 54 | 119
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 24 | 67
  Male | 2140 | 1064 | 3204
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1378 | 675 | 2053
  Not Hispanic or Latino | 804 | 413 | 1217
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 722 | 344 | 1066
  Black or African American | 584 | 301 | 885
  Other or More Than One Race | 577 | 284 | 861
  Asian | 269 | 144 | 413
  American Indian or Alaska Native | 20 | 13 | 33
  Not Collected | 8 | 2 | 10
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Puerto Rico | 9 | 2 | 11
  Argentina | 161 | 64 | 225
  United States | 431 | 233 | 664
  Brazil | 769 | 396 | 1165
  South Africa | 246 | 112 | 358
  Mexico | 8 | 4 | 12
  Thailand | 250 | 139 | 389
  Peru | 309 | 138 | 447

OUTCOME MEASURES:

1. Primary Outcome: Incidence Phase: Recent Infection Testing Algorithm (RITA) Estimate of the Background Human Immunodeficiency-1 Virus Infection Incidence Rate (bHIV) Per 100 Person Years (PY)
Description: bHIV per 100 PY in the Incidence Phase was calculated using RITA. The RITA incorporated HIV-1 testing results and recency assay testing results to estimate the bHIV. Recency assay testing was performed for participants in the All Screened Set found to have HIV-1 infection at the Incidence Phase Screening Visit as defined below. Participants were considered to have recent HIV-1 infection if the normalized optical density (ODn) was below 1.5 threshold using the Sedia limiting antigen avidity enzyme immunoassay (LAg-EIA) and the HIV-1 RNA (viral load) was > 75 copies/mL of blood.
  HIV-1 infection was defined as participants having at least one of the following central lab results at the Incidence Phase screening visit:
  * Positive HIV-1/2 differentiation Ab, OR
  * Positive HIV-1 ribonucleic acid (RNA) qualitative test, OR
  * HIV-1 RNA quantitative test ≥200 copies/mL.
Time Frame: Incidence Phase Screening Visit (Day 1)
Population: Participants in the All Screened Set were analyzed. The All Screened Set included all participants who were screened for HIV-1 in the Incidence Phase and had a non-missing HIV-1 diagnosis based on HIV test results at Incidence Phase screening. As the outcome measure was assessed prior to Randomized Blinded Phase, the data is reported in one arm consisting of all participants screened in Incidence Phase.
Measure: Number (95% Confidence Interval); unit: HIV-1 events per 100 person-years
Groups:
- Incidence Phase: All Screened Participants With Non-missing HIV-1 Diagnosis: Participants screened for HIV-1 infection and having a non-missing HIV-1 diagnosis based on results of HIV testing conducted at Incidence Phase screening.
Arm/Group | Incidence Phase: All Screened Participants With Non-missing HIV-1 Diagnosis
Number analyzed (Participants) | 4634
HIV-1 events per 100 person-years | 2.374 [1.649 to 3.417]

2. Primary Outcome: Randomized Blinded Phase: HIV-1 Incidence Reported Per 100 PY for LEN Compared to Background HIV (bHIV, Participants in All Screened Set)
Description: HIV-1 incidence per 100 PY for LEN was calculated as the number of participants who acquired HIV-1 divided by the total of a) for participants not diagnosed with HIV-1, sum of all duration of follow-up time in years, while at risk of HIV-1 infection (where a year is 365.25 days) and b) for participants diagnosed with HIV-1, sum of all duration of follow-up time up to confirmed HIV-1 diagnoses. HIV-1 diagnosis was determined by an HIV adjudication committee who reviewed potential HIV-1 infection events in the randomized participants. The committee, in a blinded, consistent, and unbiased manner, determined whether HIV test results confirmed HIV-1 infection and determined the date of diagnosis for each case, defined as the date of the earliest study visit with evidence of HIV infection considering both prospective HIV testing and back-testing of archived samples. bHIV incidence per 100 PY in All Screened Set was estimated as described in outcome measure#1.
Time Frame: Up to 149 weeks
Population: Participants in the LEN group in the Full Analysis Set (FAS) were analyzed. The FAS included all randomized participants who received at least 1 dose of any study drug and had not been diagnosed with HIV-1 on or prior to the first dose date. Per prespecified analysis, HIV-1 incidence for this outcome measure was reported only for participants who received LEN. The HIV-1 incidence was compared with participants in the All Screened Set.
Measure: Number (95% Confidence Interval); unit: HIV-1 events per 100 person-years
Arm/Group | Randomized Blinded Phase: LEN + Placebo-to-match (PTM) F/TDF | Incidence Phase: All Screened Participants With Non-missing HIV-1 Diagnosis
Number analyzed (Participants) | 2179 | 4634
HIV-1 events per 100 person-years | 0.103 [0.012 to 0.373] | 2.374 [1.649 to 3.417]
Statistical Analysis 1: Comparison: Randomized Blinded Phase: LEN + Placebo-to-match (PTM) F/TDF vs Incidence Phase: All Screened Participants With Non-missing HIV-1 Diagnosis; Null Hypothesis 01: LEN/bHIV>= 1; Null hypothesis was to be rejected if HIV-1 incidence in LEN was significantly lower than bHIV; Test type: Superiority; p < 0.0001, Wald test — p-value for rate ratio vs bHIV is from Wald test; Rate Ratio = 0.043, 95% CI 2-sided [0.010 to 0.182] — Confidence Interval (CI) for rate ratio vs bHIV is based on the delta method
Statistical Analysis 2: Comparison: Randomized Blinded Phase: LEN + Placebo-to-match (PTM) F/TDF vs Incidence Phase: All Screened Participants With Non-missing HIV-1 Diagnosis; Null Hypothesis 02: LEN/bHIV>= 0.8; Null hypothesis was to be rejected if HIV-1 incidence in LEN was significantly and at least 20% lower than bHIV; Test type: Superiority; p < 0.0001, Wald test — p-value for rate ratio vs bHIV is from Wald test; Rate Ratio = 0.043, 95% CI 2-sided [0.010 to 0.182] — CI for rate ratio vs bHIV is based on the delta method

3. Secondary Outcome: Randomized Blinded Phase: HIV-1 Incidence Reported Per 100 PY for LEN Compared to F/TDF
Description: HIV-1 incidence per 100 PY was calculated as the number of participants who acquired HIV-1 divided by the total of a) for participants not diagnosed with HIV-1, sum of all duration of follow-up time in years, while at risk of HIV-1 infection (where a year is 365.25 days) and b) for participants diagnosed with HIV-1, sum of all duration of follow-up time up to confirmed HIV-1 diagnoses. HIV-1 diagnosis was determined by an HIV adjudication committee who reviewed potential HIV-1 infection events in the randomized participants. The committee, in a blinded, consistent, and unbiased manner, determined whether HIV test results confirmed HIV-1 infection and determined the date of diagnosis for each case, defined as the date of the earliest study visit with evidence of HIV infection considering both prospective HIV testing and back-testing of archived samples.
Time Frame: Up to 149 weeks
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: HIV-1 events per 100 person-years
Arm/Group | Randomized Blinded Phase: LEN + Placebo-to-match (PTM) F/TDF | Randomized Blinded Phase: Placebo LEN + F/TDF
Number analyzed (Participants) | 2179 | 1086
HIV-1 events per 100 person-years | 0.103 [0.012 to 0.373] | 0.931 [0.426 to 1.768]
Statistical Analysis 1: Comparison: Randomized Blinded Phase: LEN + Placebo-to-match (PTM) F/TDF vs Randomized Blinded Phase: Placebo LEN + F/TDF; Test type: Other — Null Hypothesis 03: LEN - F/TDF>= 0.8/100PY; Null hypothesis was to be rejected if HIV-1 incidence in LEN is not substantially greater than F/TDF (LEN is comparable to F/TDF); p < 0.0001, Hybrid approach — p-value for rate difference (SC LEN minus F/TDF) is based on a hybrid approach; Rate difference = -0.828, 95% CI 2-sided [-1.669 to -0.255] — Exact CI for rate difference versus F/TDF is based on a hybrid approach
Statistical Analysis 2: Comparison: Randomized Blinded Phase: LEN + Placebo-to-match (PTM) F/TDF vs Randomized Blinded Phase: Placebo LEN + F/TDF; Null Hypothesis 04: LEN vs F/TDF>= 1; Null hypothesis was to be rejected if HIV-1 incidence in LEN was significantly lower than F/TDF; Test type: Superiority; p = 0.00245, Poisson model — P-value for rate ratio versus F/TDF is from a Poisson model; Rate Ratio = 0.111, 95% CI 2-sided [0.024 to 0.513] — Confidence interval for rate ratio versus F/TDF is from a Poisson model

4. Secondary Outcome: Randomized Blinded Phase: HIV-1 Incidence Among Participants Adherent to LEN
Description: A participant was defined as adherent to LEN if they have received all per-protocol administrations of LEN within 28 weeks since the previous administration. The incidence of HIV-1 infection per 100 PY calculation is defined in outcome measure #2.
Time Frame: Up to 149 weeks
Population: Participants in the Full Analysis Set who were adherent to LEN were analyzed.
Measure: Number (95% Confidence Interval); unit: HIV-1 events per 100 person-years
Arm/Group | Randomized Blinded Phase: LEN + Placebo-to-match (PTM) F/TDF
Number analyzed (Participants) | 1948
HIV-1 events per 100 person-years | 0.125 [0.015 to 0.452]

5. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs were defined as 1 or both of the following:
  Any adverse events (AEs) leading to premature discontinuation of study drug, or Any AEs with an onset date on or after the study drug start date and no later than the last exposure date after permanent discontinuation of the study drug.
  An AE was any untoward medical occurrence in a clinical study participant administered a study drug that did not necessarily have a causal relationship with the treatment.
Time Frame: Up to 4 years
Reporting Status: Not Posted

6. Secondary Outcome: Percentage of Participants Experiencing Clinically Significant Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities were defined as values that increased at least 1 toxicity grade from baseline at any post-baseline visit, up to and including the last exposure date for participants who permanently discontinued study drug, or the last available date in the database snapshot for participants who were still on treatment at the time of an analysis.
Time Frame: Up to 4 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All-Cause Mortality and Adverse Events: Up to 149 weeks
Description: All-cause Mortality: The All Randomized Analysis Set included all participants who were randomized in the study.
  Adverse Events: The Randomized Blinded Phase Safety Analysis Set included all participants who received at least 1 dose of any study drug.
Groups:
- Randomized Blinded Phase: LEN + Placebo-to-match (PTM) F/TDF: Participants received lenacapavir (LEN) 927 mg subcutaneous (SC) injection, every 26 weeks, starting on Day 1 up to for approximately 52 weeks. Participants also received loading dose of LEN 600 mg tablet orally, once daily on Day 1 and Day 2. Participants received placebo to match (PTM) emtricitabine/tenofovir disoproxil fumarate (F/TDF) tablet orally, once daily, up to approximately 52 weeks.
- Randomized Blinded Phase: Placebo LEN + F/TDF: Participants received F/TDF tablet on Day 1 orally, once daily up to for approximately 52 weeks. Participants also received PTM LEN SC injection every 26 weeks starting on Day 1 up to approximately 52 weeks and PTM LEN tablet, orally, once daily on Day 1 and Day 2.
Arm/Group | Randomized Blinded Phase: LEN + Placebo-to-match (PTM) F/TDF | Randomized Blinded Phase: Placebo LEN + F/TDF
All-Cause Mortality (participants affected / at risk) | 4/2195 | 2/1097
Serious Adverse Events (participants affected / at risk) | 71/2183 | 43/1088
Other Adverse Events (participants affected / at risk) | 1912/2183 | 882/1088
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized Blinded Phase: LEN + Placebo-to-match (PTM) F/TDF (N=2183) | Randomized Blinded Phase: Placebo LEN + F/TDF (N=1088)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Thyrotoxic periodic paralysis (Endocrine disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Strangulated umbilical hernia (Gastrointestinal disorders) | 1 | 0
Death, not otherwise specified (General disorders) | 1 | 1
Ill-defined disorder (General disorders) | 0 | 1
Lithiasis (General disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Abdominal infection (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 3 | 0
Anal abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 7 | 6
Bacterial infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0
Complicated appendicitis (Infections and infestations) | 1 | 0
Dengue fever (Infections and infestations) | 1 | 0
Dengue haemorrhagic fever (Infections and infestations) | 2 | 0
Encephalitis viral (Infections and infestations) | 1 | 0
Enteritis infectious (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Hepatitis A (Infections and infestations) | 3 | 1
Large intestine infection (Infections and infestations) | 0 | 1
Meningoencephalitis viral (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 1
Peritonsillar abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Tonsillitis bacterial (Infections and infestations) | 1 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 1
Craniofacial fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Foreign body aspiration (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound necrosis (Injury, poisoning and procedural complications) | 0 | 1
Transaminases abnormal (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Seizure (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 2
Completed suicide (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 3 | 1
Depression suicidal (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 2
Mental disorder (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0
Schizophrenia (Psychiatric disorders) | 0 | 1
Substance dependence (Psychiatric disorders) | 0 | 1
Substance use disorder (Psychiatric disorders) | 1 | 0
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 3 | 4
Suicide attempt (Psychiatric disorders) | 7 | 3
Nephrolithiasis (Renal and urinary disorders) | 1 | 1
Ureteric stenosis (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Testicular mass (Reproductive system and breast disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cellulite (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized Blinded Phase: LEN + Placebo-to-match (PTM) F/TDF (N=2183) | Randomized Blinded Phase: Placebo LEN + F/TDF (N=1088)
Diarrhoea (Gastrointestinal disorders) | 146 | 75
Nausea (Gastrointestinal disorders) | 89 | 67
Injection site erythema (General disorders) | 377 | 211
Injection site induration (General disorders) | 342 | 110
Injection site nodule (General disorders) | 1383 | 427
Injection site pain (General disorders) | 1231 | 581
Injection site swelling (General disorders) | 149 | 104
Anal chlamydia infection (Infections and infestations) | 289 | 128
Anal gonococcal infection (Infections and infestations) | 233 | 99
Influenza (Infections and infestations) | 120 | 66
Latent syphilis (Infections and infestations) | 114 | 44
Oropharyngeal gonococcal infection (Infections and infestations) | 283 | 119
Upper respiratory tract infection (Infections and infestations) | 148 | 77
Headache (Nervous system disorders) | 119 | 76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2024-10-21): https://cdn.clinicaltrials.gov/large-docs/52/NCT04925752/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-20): https://cdn.clinicaltrials.gov/large-docs/52/NCT04925752/SAP_001.pdf